CLINICAL TRIAL: NCT04048993
Title: Registry-based Biobank Development and Integrative Physiological Analysis
Status: Recruiting | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Other Study IDs: BIO
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Integrative Human Physiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Muscle biopsies, fat biopsies, microdialysate, urine, plasma, blood, dried blood spots
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Biobank development and integrative physiological analysis — Collection of biological samples (blood, urine, interstitial fluid, adipose tissue and muscle) from subjects enrolled in the Section registry, using multivariate and data-mining approaches that includes also clinical and demographic parameters.

SUMMARY:
The purpose is to develop a registry-based biobank for integrative physiological analysis based on biological samples (blood, urine, interstitial fluid and muscle) from subjects enrolled in the Section registry, using multivariate and data-mining approaches that includes also clinical and demographic parameters

ELIGIBILITY:
Inclusion Criteria:

* able to perform fatiguing exercise

Exclusion Criteria:

* severe mental or physical handicap
* chronic disease deemed by the M.D. to preclude inclusion
* use of prescription medicine deemed by the M.D. to preclude inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Human subjects able to perform exercise
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2028-08-10 (Estimated); Study Completion 2028-08-10 (Estimated)

PRIMARY OUTCOMES:
Biobank creation | through study completion, an average of 5 years
  Collection of biological samples from subjects included in the Section Registry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided